CLINICAL TRIAL: NCT00149838
Title: Optimization of Transcranial Magnetic Stimulation (TMS) for Depression
Brief Title: Magnetic Brain Stimulation for the Treatment of Adult Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH069887 (NIH); R01MH069887 (NIH); DATR A5-ETMA (Other: NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Depression
Keywords: Electric Stimulation; Magnetic Stimulation; Prefrontal Cortex; Brain
MeSH Terms: conditions — Depression | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active prefrontal rTMS phase1 (Experimental): Phase I participants receiving rTMS
  Interventions: Procedure: Prefrontal rTMS
- Sham rTMS phase 1 (Placebo Comparator): Phase I participants receiving sham stimulation
  Interventions: Procedure: Sham Stimulation
- rTMS extension (Experimental): rTMS. Phase II participants, all of whom did not meet remission requirements after phase 1. They all receive active open label rTMS
  Interventions: Procedure: Prefrontal rTMS
- Open label antidepressant regimen (Experimental): All patients who met remission who were then transitioned to medications after the TMS trial was completed.
  Interventions: Drug: Antidepressant Regimen

INTERVENTIONS:
Procedure: Prefrontal rTMS — Participants receive 120% motor threshold (MT) over left and right prefrontal cortex. Treatments will be administered daily for 3 weeks. Participants who show signs of improvement may continue Phase I for up to 3 additional weeks.
  Other Names: TMS; rTMS
  Arms: Active prefrontal rTMS phase1; rTMS extension
Drug: Antidepressant Regimen — Particpants who acheive remission with rTMS may start antidepressant medication in phase III.
  Other Names: medication
  Arms: Open label antidepressant regimen
Procedure: Sham Stimulation — The sham stimulation will mimic the sensation of rTMS but will not induce an intracerebral current. Treatments will be administered daily for 3 weeks.
  Arms: Sham rTMS phase 1

SUMMARY:
This study will evaluate the safety and effectiveness of magnetic brain stimulation for the treatment of major depression in depressed adults with moderate treatment resistance.

DETAILED DESCRIPTION:
Major depression is a type of depression that can interfere with the ability to work, study, sleep, eat, and enjoy once pleasurable activities. Because people often develop resistances to medications used to treat depression, new treatments are needed. Decreased electrical activity in the prefrontal region of the brain has been linked to some symptoms of depression. Repetitive transcranial magnetic stimulation (rTMS) can be used to influence the brain's electrical activity. This procedure entails attaching electrodes to the head and using a device to pass magnetic energy through coils and into the brain. rTMS has been shown to have antidepressant effects in depressed individuals. However, optimal levels of intensity and treatment duration have yet to be determined. This study will assess the safety and effectiveness of rTMS on the prefrontal region of the brain in depressed adults with moderate treatment resistance.

The treatment phase of this double-blind study will last a minimum of 32 weeks and will consist of 3 phases. In Phase I, participants will be randomly assigned to receive either rTMS or sham stimulation. The sham stimulation will mimic the sensation of rTMS but will not induce an intracerebral current. Treatments will be administered daily for 3 weeks. Participants who show signs of improvement may continue Phase I for up to 3 additional weeks. In Phase II, participants who were unresponsive to Phase I treatment will receive daily rTMS at a lower dose for 3 weeks. Participants who show signs of improvement, but have not achieved remission, may continue Phase II for 4 additional weeks. Baseline magnetic resonance images will be used to determine the optimal stimulus intensity by adjusting for individual differences in cortical to skull distances. Phase III participants will be only those who achieved remission in the first 2 phases. These participants will receive antidepressant medication treatment daily for six months. Participants' functional status and symptoms of depression will be measured using self-report scales and video-recorded interviews at study start date and at the end of each treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression with a current episode
* Hamilton Rating Scale for Depression score higher than 20
* No response or intolerance to antidepressant medication in the current depressive episode

Exclusion Criteria:

* Current use of antidepressants
* Diagnosis of psychosis or anxiety disorder
* Current substance abuse
* Seizures or history of head trauma

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2005-02; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. George, MD, Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Columbia University, New York, New York
  - Brain Stimulation Laboratory, Medical University of South Carolina, Charleston, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers can email the PI, Dr. George, with a request and how they plan to analyze the data. He will then make available a de-identified copy of the data.

REFERENCES:
- [Derived] Borckardt JJ, Nahas ZH, Teal J, Lisanby SH, McDonald WM, Avery D, Durkalski V, Pavlicova M, Long JM, Sackeim HA, George MS. The painfulness of active, but not sham, transcranial magnetic stimulation decreases rapidly over time: results from the double-blind phase of the OPT-TMS Trial. Brain Stimul. 2013 Nov;6(6):925-8. doi: 10.1016/j.brs.2013.04.009. Epub 2013 May 21. PMID 23769413
- [Derived] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TMS: Phase I participants receiving rTMS
  Prefrontal Repetitive Transcranial Magnetic Stimulation (rTMS): Participants receive 120% motor threshold (MT) over left and right prefrontal cortex. Treatments will be administered daily for 3 weeks. Participants who show signs of improvement may continue Phase I for up to 3 additional weeks.
- Sham TMS: Phase I participants receiving sham stimulation
  Sham Stimulation: The sham stimulation will mimic the sensation of rTMS but will not induce an intracerebral current. Treatments will be administered daily for 3 weeks.
- rTMS Extension: Phase II participants, all of whom did not meet remission requirements after phase 1. They will all receive active open label rTMS
Period: Phase I
Arm/Group | Active TMS | Sham TMS | rTMS Extension | Open Label Antidepressant Regimen
Started | 92 | 98 | 0 | 0
Completed | 72 | 82 | 0 | 0
Not Completed | 20 | 16 | 0 | 0
Period: Phase II
Arm/Group | Active TMS | Sham TMS | rTMS Extension | Open Label Antidepressant Regimen
Started | 0 | 0 | 144 | 0
Completed | 0 | 0 | 144 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase III
Arm/Group | Active TMS | Sham TMS | rTMS Extension | Open Label Antidepressant Regimen
Started | 0 | 0 | 0 | 61
Completed | 0 | 0 | 0 | 37
Not Completed | 0 | 0 | 0 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 92 | 98 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.6) | 46.5 (12.3) | 47.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 105
  Male | 37 | 48 | 85

OUTCOME MEASURES:

1. Primary Outcome: Depression Remission, as Measured by the Hamilton Rating Scale for Depression
Description: The Hamilton Rating Scale for Depression 17-item total score ranges from 0 to 52 with higher scores indicating more depression. Remission is defined as a total score of ≤ 8
Time Frame: Measured at the end of Phases 1, 2, and 3
Population: Remission
Measure: Number; unit: number of remitted patients
Groups:
- Active Open for 3 Weeks: Phase II participants
  Lower Dose rTMS: Participants who are unresponsive to Phase I treatment with rTMS will continue a lower dose of rTMS for an additional 3 to 7 weeks in Phase II.
- Medication Followup: Phase III participants
  Antidepressant Regimen: Particpants who acheive remission with rTMS may start antidepressant medication in phase III.
Arm/Group | Active TMS | Sham TMS | Active Open for 3 Weeks | Medication Followup
Number analyzed (Participants) | 92 | 98 | 141 | 55
number of remitted patients | 13 | 5 | 43 | 12

ADVERSE EVENTS:
Groups:
- rTMS Extension: rTMS. Phase II participants, all of whom did not meet remission requirements after phase I. They all receive active open label rTMS
Arm/Group | Active TMS | Sham TMS | rTMS Extension | Open Label Antidepressant Regimen
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/98 | 0/144 | 0/61
Other Adverse Events (participants affected / at risk) | 18/92 | 15/98 | 0/144 | 0/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=92) | Sham TMS (N=98) | rTMS Extension (N=144) | Open Label Antidepressant Regimen (N=61)
All adverse events (Psychiatric disorders) | 18 (18) | 15 (15) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No